CLINICAL TRIAL: NCT06783530
Title: Psychological and Clinical Outcomes After Splint Therapy with Versus Without Doctor-patient Communication Concept in the Management of TMDs
Brief Title: Psychological and Clinical Outcomes of Splint Therapy with and Without Doctor-Patient Communication in TMD Management
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soaad Tolba Mohammed Tolba Badawi (Other)
Responsible Party: Sponsor-Investigator, Soaad Tolba Mohammed Tolba Badawi, lecturer of oral and maxillofacial department, faculty of dentistry, Mansoura university, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02012024OS
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Disorders (TMDs)
Keywords: Splint Therapy; Doctor-Patient Communication; Non-Surgical TMD Treatment; TMDs management
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model with two groups: one receiving standard splint therapy and the other receiving splint therapy with enhanced doctor-patient communication.
Who Masked: Participant, Outcomes Assessor
Masking Description: The allocation was concealed from participants and the statistician performing the data analysis to minimize bias. However, the clinician administering the intervention was aware of the patient's allocation to ensure appropriate treatment delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Splint Therapy with Enhanced Doctor-Patient Communication (Experimental): Participants in this arm received splint therapy along with structured doctor-patient communication to improve treatment outcomes.
  Interventions: Behavioral: Splint Therapy with Enhanced Doctor-Patient Communication
- Standard Splint Therapy (Active Comparator): Participants in this group received standard splint therapy for the management of temporomandibular disorders (TMD). The splint was fitted and adjusted by a qualified clinician, and participants was monitored for outcomes such as pain reduction, jaw function, and patient satisfaction.
  Interventions: Device: Splint Therapy

INTERVENTIONS:
Behavioral: Splint Therapy with Enhanced Doctor-Patient Communication — A structured communication protocol aimed at improving doctor-patient interaction and treatment adherence.
  Arms: Splint Therapy with Enhanced Doctor-Patient Communication
Device: Splint Therapy — A custom-fitted occlusal splint designed to alleviate symptoms of temporomandibular disorders (TMD).
  Arms: Standard Splint Therapy

SUMMARY:
This study aimed to evaluate the psychological and clinical outcomes of patients undergoing splint therapy with or without enhanced doctor-patient communication in the management of temporomandibular disorders (TMDs). The study compared treatment approaches to determine their impact on patient satisfaction and clinical results.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMDs) are prevalent conditions characterized by jaw pain, functional limitations, and psychological distress. This study investigated the impact of splint therapy combined with enhanced doctor-patient communication on psychological well-being and clinical outcomes. Participants were randomly assigned to receive standard splint therapy or splint therapy with additional doctor-patient communication strategies. The primary outcomes include clinical and psychological status improvements, measured over six months, and patient satisfaction, assessed over a one-year period. The results aimed to provide insights into optimizing treatment strategies for TMD patients.

ELIGIBILITY:
Inclusion Criteria:

* patients complaining of pain in the orofacial region (either arthrogenous and/or myogenous TMD) in the last 3 months, who never underwent any type of treatment for TMD's.
* Age ≥16 years.

Exclusion Criteria:

* patients who have already undergone any treatment for TMD's, edentulous patients,
* patients with any systemic disease that could cause joint and/or muscle changes,
* patients who were undergoing drug treatment for the condition, current pregnancy, or breastfeeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress levels | Baseline to 6 months.
  Depression, anxiety, and stress levels was measured using the 10-item Depression, Anxiety, and Stress Scale (DASS-10) at baseline and after six months of therapy. The DASS-10 comprises 10 items, each rated on a 4-point Likert scale ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much or most of the time").
  * Minimum value: 0
  * Maximum value: 30
  * Interpretation: Higher scores indicate worse psychological outcomes.
Change in Interincisal Mouth Opening | Baseline to 6 months.
  Maximum interincisal mouth opening was measured at baseline and after six months of therapy using a calibrated caliper.
Change in Intra-articular pain (IAP) | Baseline to 6 months.
  Intra-articular pain was assessed at baseline and after six months using the Visual Analog Scale (VAS) for pain intensity. The scale ranged from 0 to 10, where:
  * Minimum value: 0 (No pain)
  * Maximum value: 10 (Worst possible pain).
Change in Joint Sound Presence and Characteristics | Baseline to 6 months.
  Joint Sounds were measured in scores from 0 to 5, where 0 = no joint sound, 1 = Joint noise on occasion, 2 = palpable clicking, 3 = audible clicking, 4 = absence of previous clicking (closed lock), and 5 = crepitation. Assessment of the presence and characteristics of joint sounds was performed at baseline and after six months of therapy.

SECONDARY OUTCOMES:
Change in Masticatory Muscle Pain Intensity | Baseline to 6 months.
  Pain intensity in the masticatory muscles (e.g., masseter, temporalis, medial pterygoid, lateral pterygoid) was assessed by palpation at specific points, which uses a pain scale from zero to three (0: pressure only; 1: mild pain; 2: moderate pain; 3: severe pain). Pain assisted by palpation pressure (1kg pressure for 5sec) as defined in DC/TMD.
Patient Satisfaction with Treatment | From 6 months to 1-year post-intervention.
  Each patient was evaluated at 6 and 12 months after intervention. The patient satisfaction questionnaire comprised two questions assessed using a 10-point Likert scale (1 = extremely dissatisfied to 10 = perfect/strongly satisfied).
  * Overall satisfaction with the clinical result of the treatment.
  * Satisfaction with the fulfillment of postoperative expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Soaad Tolba Badawy, Lecturer of OMFS, MU, Principal Investigator — Faculty of dentistry, Mansoura university; Mai Ahmed Haggag, Assistant Professor of OMFS, Principal Investigator — Faculty of dentistry, Mansoura university; Christine Raouf Micheal, Assistant Professor, Principal Investigator — Prosthodontics Department, Faculty of dentistry, Mansoura university
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no decision has been made regarding the sharing of Individual Participant Data (IPD). Data-sharing plans will be determined based on institutional guidelines, ethical considerations, and journal requirements at the time of publication.

REFERENCES:
- [Background] de Barros Pascoal AL, de Freitas RFCP, da Silva LFG, Oliveira AGRC, Dos Santos Calderon P. Effectiveness of Counseling on Chronic Pain Management in Patients with Temporomandibular Disorders. J Oral Facial Pain Headache. 2020 Winter;34(1):77-82. doi: 10.11607/ofph.2163. Epub 2019 Apr 12. PMID 30978270
- [Derived] Haggag MA, Ibrahim CRM, Badawy ST. Psychological and Clinical Outcomes After Splint Therapy With Versus Without Doctor-Patient Communication Concept in the Management of TMDs: A Randomised Controlled Clinical Trial. J Oral Rehabil. 2025 Oct;52(10):1651-1663. doi: 10.1111/joor.14005. Epub 2025 May 19. PMID 40384540
- See also: This link provides a collection of research articles related to splint therapy for temporomandibular disorders, which aligns with the focus of this study. — https://pubmed.ncbi.nlm.nih.gov/?term=splint+therapy+for+temporomandibular+disorders.%22
- See also: This link directs to a PubMed search for studies related to counselling as a treatment approach for temporomandibular disorders, which is relevant to this study's objectives. — https://pubmed.ncbi.nlm.nih.gov/?term=counselling+for+temporomandibular+disorders.%22
- Available data/document: Study Protocol — https://dentfac.mans.edu.eg — Faculty of Dentistry, Mansoura University - Ethical Committee Information.